CLINICAL TRIAL: NCT02568124
Title: Tranexamic Acid in Chronic Subdural Hematomas
Acronym: TRACS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Dr David Mathieu, M.D., Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-213
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Chronic Subdural Hematoma
Keywords: Tranexamic acid; Cyklokapron; Conservative management; Medical management
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Experimental): Tranexamic acid 750 mg daily until complete radiological resolution of the chronic subdural hematoma or a maximum of 20 weeks.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Placebo tablet daily until complete radiological resolution of the chronic subdural hematoma or a maximum of 20 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Other Names: Cyklokapron
  Arms: Tranexamic acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
BACKGROUND Chronic subdural hematoma (CSDH) is one of the most frequent reasons for cranial neurosurgical consult. There is no widely accepted medical treatment for CSDH.

This trial will investigate whether Tranexamic Acid (TXA) can increase the rate of CSDH resolution following conservative management, lower the number of required surgical procedures and decrease the rate of CSDH recurrence following surgical evacuation. TRACS is a double blind, randomized, parallel-design, placebo-controlled, phase IIB study designed to provide preliminary efficacy data as well as feasibility, safety and incidence data required to plan a larger definitive phase III trial.

METHODS Consecutive patients presenting at the Centre Hospitalier Universitaire de Sherbrooke with a recent (< 14 days) diagnosis of subdural hematoma with a chronic component will be screened for eligibility. Exclusion criteria include specific risk factors for thromboembolic disease, anticoagulant use or contraindication to TXA. A total of 130 patients will be randomized to receive either 750 mg of TXA daily or placebo until complete radiological resolution of the CSDH or for a maximum of 20 weeks. CSDH volume will be measured on serial CT scanning. Cognitive function tests, quality of life questionnaires as well as functional autonomy assessments will be performed at enrollment, 10 weeks follow-up and 3 months post-treatment follow-up. During the treatment period, patients will undergo standard CSDH management with surgery being performed at the discretion of the treating physician. If surgery is performed, the CSDH and its outer membrane will be sampled for in vitro analysis.

The primary outcome is the rate of CSDH resolution at 20 weeks without intervening unplanned surgical procedure. Secondary outcomes include CSDH volume, incidence of surgical evacuation procedures, CSDH recurrence, cognitive functions, functional autonomy, quality of life, incidence of complications and length of hospital stay. Planned subgroup analyses will be performed for conservatively vs surgically-managed subjects and highly vs poorly vascularised CSDH.

DISCUSSION CSDH is a frequent and morbid condition for which an effective medical treatment has yet to be discovered. The TRACS trial will be the first prospective study of TXA for CSDH.

ELIGIBILITY:
Inclusion Criteria:

* CT scan demonstrating the existence of a subdural hematoma containing a chronic component
* Diagnosis within the last 14 days

Exclusion Criteria:

* Acute subdural hematoma with no chronic component;
* Active thrombotic, thromboembolic or atheroembolic disease, including deep venous thrombosis within the last six months, cerebral thrombosis within the last six months, symptomatic carotid stenosis who did not undergo surgery or stroke within the last year;
* Past history of unprovoked deep venous thrombosis or idiopathic pulmonary embolism;
* Known hereditary thrombophilia, including Factor V Leiden, Antithrombin III mutation, Protein C deficiency, Protein S deficiency;
* Atrial fibrillation (unless under successful rhythm control therapy);
* Metallic heart valve;
* Vascular stenting procedure within the last year;
* Cardiac or vascular surgical procedure within the last 6 months, including endarterectomy, bypass or angioplasty;
* Ongoing investigation for suspected malignancy;
* Confirmed active malignancy;
* Concomitant hormone therapy for malignancy;
* Concomitant hormone contraceptive pill;
* Macroscopic hematuria;
* Known or suspected tranexamic acid allergy;
* Pregnancy or breastfeeding;
* Concomitant use of anticoagulant medication;
* Any concern from the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-11; Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Hematoma resolution | 20 weeks
  The rate of chronic subdural hematoma resolution without intervening unplanned surgical procedure. Specifically, if the initial management strategy chosen by the attending physician within the first 24 hours of presentation consists of expectant management, any surgical procedure leads to a failure of meeting the primary outcome. On the other hand, if the management strategy chosen by the attending physician within the first 24 hours of presentation included a surgical evacuation of the CSDH, the primary outcome is met if the control CT scan at 20 weeks demonstrates a complete radiological resolution of the CSDH. Should a second surgery be required, the subject will fail to meet the primary outcome even if the CSDH has completely resolved by 20 weeks.

SECONDARY OUTCOMES:
Hematoma volume | 20 weeks
  Measured by segmentation analysis on the 20 weeks CT scan
Surgical evacuation | 32 weeks
  The incidence of surgical evacuation procedures
Hematoma recurrence | 32 weeks
Cognitive function | 10 weeks
  Assessed by the Montreal Cognitive Assessment (MoCA) and Mini-Mental State Examination (MMSE)
Cognitive function | 32 weeks
  Assessed by the Montreal Cognitive Assessment (MoCA) and Mini-Mental State Examination (MMSE)
Functional autonomy | 10 weeks
  Assessed by the modified Barthel Index (mBI) and Glasgow Outcome Scale Extended (GOSE)
Functional autonomy | 32 weeks
  Assessed by the modified Barthel Index (mBI) and Glasgow Outcome Scale Extended (GOSE)
Quality of life scores at 10 weeks | 10 weeks
  Assessed by the EQ-5D-5L and the Sherbrooke Neuro-oncology Assessment Scale (SNAS)
Quality of life scores at 32 weeks | 32 weeks
  Assessed by the EQ-5D-5L and the Sherbrooke Neuro-oncology Assessment Scale (SNAS)
Length initial of hospital stay | 32 weeks
Number of rehospitalisation | 32 weeks
Complications | 32 weeks
  Incidence of any complication related to tranexamic acid administration

CONTACTS AND LOCATIONS:
Overall Officials: David Mathieu, M.D., Principal Investigator — Université de Sherbrooke
Locations (3):
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre Hospitalier Affilié Universitaire de Québec, Québec

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Iorio-Morin C, Blanchard J, Richer M, Mathieu D. Tranexamic Acid in Chronic Subdural Hematomas (TRACS): study protocol for a randomized controlled trial. Trials. 2016 May 5;17(1):235. doi: 10.1186/s13063-016-1358-5. PMID 27150916